CLINICAL TRIAL: NCT04658836
Title: Triamcinolone Acetonide Levels in Cochlear Perilymph, Lateral Canal and CSF in Patients With Vestibular Schwannomas
Brief Title: Triamcinolone Levels in Cochlear Perilymph, Lateral Canal and CSF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christoph Arnoldner, Principal Investigator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TACCSF
Record Dates: First submitted 2020-06-23; First posted 2020-12-09 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Vestibular Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triamcinolone application (Experimental): Patients will recieve intratympanic triamcinolone acetonide 24h before vestibular schwannoma surgery
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40mg/mL — Intratympanic application of triamcinolone acetonide

SUMMARY:
Patients undergoing surgery of a vestibular schwannoma will be included in the study. Patients will receive triamcinolone acetonide 24h before surgery. During translabyrinthine surgery cochlear perilymph, perilymph from the semicircular canal and cerebrospinal fluid will be taken and analyzed for triamcinolone content. In patients undergoing middle fossa or retrosigmoid resection only cerebrospinal fluid will be taken and analyzed for triamcinolone acetonide level.

DETAILED DESCRIPTION:
Patients between 18 and 90 years undergoing surgery of a vestibular schwannoma will be included in the study. Patients will be offered an application of triamcinolone acetonide intratympanically on the day before surgery.

During surgery samples will be taken to define how much triamcinolone acetonide enters into the perilymphatic fluid, the perilymph of the semicircular canals and CSF.

Patients undergoing translabyrinthine surgery will undergoing labyrinthectomy during which samples of the semicircular canal can be taken. During translabyrinthine surgery nerve monitoring will be carried out using an intracochlear electrode. Before inserting the electrode perilymph of the cochlea can be taken. Immediately after opening the dura cerebrospinal fluid will be taken. Patients undergoing middle fossa or retrosigmoid resection of the vestibular schwannoma will not undergo sampling of the perilymph. In these patients cerebrospinal fluid will be taken to determine triamcinolone acetonide levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 90 years undergoing a surgery of the cerebellopontine angle due to vestibular schwannoma and who are willing to participate in the study

Exclusion Criteria:

* Patients younger than 18 years Patients who receive cortison regularly or receive cortison i.v. or p.o. preoperatively Patients with contraindications against the administration of VolonâA

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Triamcinolone acetonide level | one day
  Drug level

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Arnoldner, Principal Investigator — Medical University of Vienna, Otorhinolaryngology, Head and Neck Surgery
Locations (1):
- Medical University of Vienna (AKH), Vienna, Austria

IPD SHARING:
Plan to Share IPD: No